CLINICAL TRIAL: NCT06285422
Title: A Phase 1 Study Evaluating SC262, a Hypoimmune, Allogeneic CD22-directed CAR T Cell Therapy, in Relapsed and/or Refractory Non-Hodgkin's Lymphoma (VIVID)
Brief Title: Study Evaluating SC262 in Subjects With r/r Non-Hodgkin's Lymphoma (VIVID)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sana Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC262-101
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Non Hodgkin's Lymphoma; Large B-cell Lymphoma
Keywords: Large B-Cell Lymphoma; CAR T Cell Therapy; Mantle Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; High-Grade B-Cell Lymphoma; Primary Mediastinal B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma; Non-Hodgkin's Lymphoma; Allogeneic; Hypoimmune; CD22; SC262
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SC262 Plus Chemotherapy Regimen (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment with SC262
  Interventions: Drug: SC262

INTERVENTIONS:
Drug: SC262 — SC262 is an allogeneic CAR -T cell therapy
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
SC262-101 is a Phase 1 study to evaluate SC262 safety and tolerability, anti-tumor activity, cellular kinetics, immunogenicity, and exploratory biomarkers.

DETAILED DESCRIPTION:
This is an open-label, single arm, Phase 1, first-in-human (FIH) study to evaluate the safety and tolerability of SC262 administered intravenously (IV) following a standard lymphodepleting chemotherapy regimen of cyclophosphamide and fludarabine in subjects with Non Hodgkin's Lymphoma (NHL) who have received no more than 1 prior CD19-directed Chimeric Antigen Receptor T-Cells (CAR T) cell therapy. This study will be conducted in 2 parts. Dose finding using a 3+3 design in subjects with NHL. Dose expansion to further evaluate safety and efficacy at the recommended phase 2 dose (RP2D) in subjects with Large B-Cell Lymphoma (LBCL).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female Subject aged 18-80 years at the time of signing the informed consent
2. Histologic diagnosis of NHL (based on World Health Organization 2016 criteria) including:

   * LBCL, including Diffuse Large B Cell Lymphoma (DLBCL) not otherwise specified (NOS) (including DLBCL arising from indolent lymphoma), Primary Mediastinal Large B-Cell Lymphoma (PMBCL), High-Grade B-Cell Lymphoma (HGBCL), and Follicular Lymphoma (FL) Grade 3B
   * FL
   * Marginal Zone Lymphomas (MZL)
   * Mantle Cell Lymphoma (MCL)
3. Relapsed or refractory disease after no more than 1 prior CD19-directed CAR T cell therapy
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
5. At least 1 measurable (PET-positive) lesion per Lugano classification
6. Life expectancy ≥12 Weeks

Exclusion Criteria:

1. Prior CD22-directed therapy including CD22-directed CAR T cell therapy or other CD22 -directed antibody or cell therapy (e.g., Natural Killer (NK) cell)
2. History of central nervous system (CNS) involvement of lymphoma within 1 year prior to enrollment.
3. Autologous hematopoietic stem cell transplantation (HSCT) within 3 months before treatment with Lymphodepleting (LD) chemotherapy (or allogeneic HSCT at any time)
4. Active autoimmune disease or any other diseases requiring immunosuppressive therapy or corticosteroid therapy (defined as >10 mg/day prednisone or equivalent)
5. History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement, within 12 months of enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of SC262 | 24 months
  Safety and Tolerability: Proportion of subjects experiencing adverse events and dose-limiting toxicities

SECONDARY OUTCOMES:
Evaluate preliminary anti-tumor activity of SC262 | 24 months
  Preliminary anti-tumor activity: Proportion of subjects with an objective response (including partial response or complete response)
Evaluate cellular kinetics and persistence of SC262 | 24 months
  Cellular kinetics related peak (Cmax) in peripheral blood
Evaluate cellular kinetics and persistence of SC262 | 24 months
  Cellular kinetics-related parameters evaluated by CAR T cell copy number
Evaluate cellular kinetics and persistence of SC262 | 24 months
  Area under the concentration time curve (AUC) in peripheral blood
Evaluate host immunogenicity to SC262 | 24 months
  Incidence of anti-CD19-directed CAR antibodies

CONTACTS AND LOCATIONS:
Overall Officials: John Gerecitano, MD, PhD, Study Director — Sana Biotechnology, Inc.
Locations (3):
- United States (3):
  - The University of Kansas Hospital, Kansas City, Kansas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington